CLINICAL TRIAL: NCT06677359
Title: Impact of Creatine Monohydrate Micronized Supplementation With or Without Multicomponent Training in Older Adults.
Acronym: CREAGED
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundacion Miguel Servet (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: CREAGED
Record Dates: First submitted 2024-10-22; First posted 2024-11-06 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Functionality; Cognition; Strength Training Effects
Keywords: creatine; supplementation; multicomponent training; older people

STUDY DESIGN:
Intervention Model Description: Unicenter Randomized Clinical Trial
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Control group (Placebo Comparator): Participants will recieved placebo supplementation without multicomponent training intervention.
  Interventions: Dietary Supplement: Placebo Group
- Creatine group (Experimental): Participants will recieved micronized creatine monohydrate supplementation without multicomponent training intervention.
  Interventions: Dietary Supplement: Creatine Group
- Control multicomponent training group (Active Comparator): Participants will recieved placebo supplementation and multicomponent training intervention
  Interventions: Dietary Supplement: Placebo Group; Other: Multicomponent Training
- Creatine multicomponent training group (Experimental): Participants will recieved micronized creatine monohydrate supplementation and multicomponent training intervention.
  Interventions: Dietary Supplement: Creatine Group; Other: Multicomponent Training

INTERVENTIONS:
Dietary Supplement: Creatine Group — Micronized creatine monohydrate supplementation.
  Arms: Creatine group; Creatine multicomponent training group
Dietary Supplement: Placebo Group — Participants will recieved placebo supplementation
  Arms: Control group; Control multicomponent training group
Other: Multicomponent Training — Multicomponent physical exercise intervention
  Arms: Control multicomponent training group; Creatine multicomponent training group

SUMMARY:
The goal of this clinical trial is to study and evaluate whether a protocol of creatine supplementation, with or without multicomponent training, improves functional and cognitive capacity in individuals over 75 years old. The results of this study will further our understanding of creatine supplementation effects in the context of older patients and in combination with multicomponent training, thereby enhancing patient care strategies. Additionally, the goal is to improve the quality of life for the elderly and the efficiency of the healthcare system.

The main questions it aims to answer are:

1. Does creatine supplementation alone provide physical, functional and cognitive benefits to people over 75 years of age?
2. Is creatine supplementation safe for people over 75 years old?

Researchers will compare creatine monohydrate supplementation with or without multicomponent training intervention to placebo supplementation with or without multicomponent training intervention to see if the creatine supplementation protocol leads to significant improvements in functional and cognitive outcomes. This comparison will help determine the effectiveness of the supplementation intervention in enhancing the overall well-being of elderly patients.

Participants will:

* Engage in a structured multicomponent exercise program designed specifically for elderly patients. This program will include activities focused on strength training, balance exercises, and walking to improve mobility and reduce the risk of falls.
* Attend supervised exercise sessions several times a week, allowing for individualized attention and adjustments based on each participants abilities and health status.
* Be monitored for changes in functional capacity using standardized assessments, which will measure improvements in mobility, strength, and overall physical functioning.
* Undergo cognitive assessments to evaluate any changes in cognitive status throughout the intervention and during follow-up periods after discharge.
* Participate in surveys and interviews to assess their quality of life, including physical, emotional, and social well-being, before and after the intervention.
* Attend follow-up assessments at designated intervals to track their progress and outcomes, ensuring that any long-term benefits of the exercise program are recognized and documented.

Inclusion criteria will focus on individuals aged over 75 years. Participants must be capable of communication and ambulation, either independently or with assistance.

* Life expectancy ≥ 6 months.
* Barthel Index > 60.

Exclusion criteria will ensure the safety and appropriateness of the intervention. Individuals who explicitly refuse to participate or cannot provide informed consent will be excluded. Additionally, those with a life expectancy of less than three months, terminal illnesses, or significant medical contraindications for exercise will not be eligible. Participants with moderate to severe neurocognitive disorders or disabilities that severely limit mobility will also be excluded to maintain the integrity of the intervention.

This clinical trial aims to recruit a total of 120 participants from the Geriatric Department or Primary Care, providing a comprehensive dataset to analyze the effectiveness and safety of the multicomponent exercise program. By examining the outcomes related to functional capacity, cognitive status, and quality of life, the study seeks to provide valuable insights into the benefits of physical activity for elderly patients during hospitalization.

DETAILED DESCRIPTION:
The goal of this clinical trial is to study and evaluate whether a protocol of creatine supplementation, with or without multicomponent training, improves functional and cognitive capacity in individuals over 75 years old. The results of this study will further our understanding of creatine supplementation effects in the context of older patients and in combination with multicomponent training, thereby enhancing patient care strategies. Additionally, the goal is to improve the quality of life for the elderly and the efficiency of the healthcare system.

The main questions it aims to answer are:

1. Does creatine supplementation alone provide physical, functional and cognitive benefits to people over 75 years of age?
2. Is creatine supplementation safe for people over 75 years old?
3. Could the creatine supplementation does enhances benefits of multicomponent training exercise physical protocol?
4. Is the creatine supplementation time of 5 weeks sufficient to observe measurable effects in this population?

Researchers will compare creatine monohydrate supplementation with or without multicomponent training intervention to placebo supplementation with or without multicomponent training intervention to see if the creatine supplementation protocol leads to significant improvements in functional and cognitive outcomes. This comparison will help determine the effectiveness of the supplementation intervention in enhancing the overall well-being of elderly patients.

Participants will:

* Engage in a structured multicomponent exercise program designed specifically for elderly patients. This program will include activities focused on strength training, balance exercises, and walking to improve mobility and reduce the risk of falls. The exercises will be tailored to the individual capabilities of each participant, ensuring safety and effectiveness.
* Attend supervised exercise sessions several times a week, allowing for individualized attention and adjustments based on each participants abilities and health status. These sessions will be conducted by trained physical therapists who specialize in geriatric care.
* Be monitored for changes in functional capacity using standardized assessments, which will measure improvements in mobility, strength, and overall physical functioning. Assessments will include tools such as the Timed Up and Go Test (TUG) and Short Physical Performance Battery (SPPB).
* Undergo cognitive assessments to evaluate any changes in cognitive status throughout the intervention and during follow-up periods after discharge. Cognitive evaluations will include tests like the Mini-Mental State Examination (MMSE) and the Montreal Cognitive Assessment (MoCA).
* Participate in surveys and interviews to assess their quality of life, including physical, emotional, and social well-being, before and after the intervention. Quality of life will be measured using validated tools such as and the EuroQol-5D (EQ-5D).
* Attend follow-up assessments at designated intervals to track their progress and outcomes, ensuring that any middle-term benefits of the exercise program are recognized and documented. Follow-ups will occur at 5 weeks post-discharge.

Inclusion criteria will focus on individuals aged over 75 years. Participants must be capable of communication and ambulation, either independently or with assistance.

The inclusion criteria will focus on individuals aged over 75 years, also:

* Able to ambulate with or without personal/technical assistance.
* Life expectancy ≥ 6 months.
* Barthel Index > 60.
* Informed consent by patients, or legal representatives.

Exclusion criteria will ensure the safety and appropriateness of the intervention. Individuals who explicitly refuse to participate or cannot provide informed consent will be excluded. Additionally, those with a life expectancy of less than three months, terminal illnesses, or significant medical contraindications for exercise will not be eligible. Participants with moderate to severe neurocognitive disorders or disabilities that severely limit mobility will also be excluded to maintain the integrity of the intervention.

Sample Size and Recruitment: This clinical trial aims to recruit a total of 120 participants. Recruitment will be conducted through Geriatric Department or Primary Care, with potential participants identified by medical staff and referred to the research team. Informed consent will be obtained from all participants or their legal representatives prior to enrollment.

Data Collection and Analysis: Data will be collected at baseline, during the intervention, and at follow-up assessments. This will include demographic information, clinical history, baseline functional and cognitive assessments, and post-intervention evaluations. Statistical analyses will be performed to compare outcomes between the intervention and control groups, using appropriate methods to account for potential confounding factors.

Ethical Considerations: This study will adhere to ethical guidelines for research involving human subjects. The protocol will be reviewed and approved by the Institutional Review Board (IRB) at each participating center. Informed consent will be obtained from all participants, ensuring they understand the study purpose, procedures, risks, and benefits.

Expected Outcomes: The findings of this study may provide valuable insights into the impact of creatine monohydrate supplementation for elderly participants. By examining the outcomes related to functional capacity, cognitive status and quality of life, the study seeks to inform future guidelines and practices for improving the care of older adults. Additionally, the research may contribute to the understanding of how creatine supplementation can positively influence health at the molecular level, potentially leading to new therapeutic approaches for managing health in elderly populations.

ELIGIBILITY:
Inclusion Criteria:

* Age: 75 years or older.
* Able to ambulate with or without personal/technical assistance.
* Life expectancy ≥ 6 months.
* Barthel Index > 60.
* Informed consent by patients, or legal representatives.

Exclusion Criteria:

* Global Deterioration Scale (GDS 6-7).
* Intolerance or allergy foods or drugs.
* Deglutition problems (Dx: dysphagia)
* Any pathological or metabolic condition incompatible with physical exercise.
* Creatine supplementation for less than 6 weeks.
* Consumption of more than 200 mg of caffeine daily.
* Supervised physical training.

Min Age: 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-11-30 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Function | Through study completion, an average of 10 weeks
  Short Performance Physical Battery (SPPB)
Strength | Through study completion, an average of 10 weeks
  Maximus Repetition (RM)
Cognition | Through study completion, an average of 10 weeks
  Cognition Test: MMSE.

SECONDARY OUTCOMES:
Muscle Status | Through study completion, an average of 10 weeks
  Muscle ultrasound.
Security | Through study completion, an average of 10 weeks
  Glomerular filtration rate (GFR)
Anthropometrical Measurements | Through study completion, an average of 10 weeks
  Bioimpedance: PHASE ANGLE (PhA), Fat-Free Mass (FFM) and Muscle Mass (MM)

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas Martinez-Velilla, PhD, Principal Investigator — Navarrabiomed-Fundación Miguel Servet-Hospital de Navarra
Locations (1):
- Hospital Universitario de Navarra, Pamplona, Navarre, Spain